CLINICAL TRIAL: NCT02722720
Title: Prospective, Randomized, Single Center Study of Atherothrombotic and Thromboembolic Events After Carotid Artery Stenting Using Transfemoral and Transradial Approach
Brief Title: Carotid Arteries Stenting Complications: Transradial Approach Versus Transfemoral
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASTE-1.0
Record Dates: First submitted 2016-03-13; First posted 2016-03-30 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Carotid Atherosclerosis; Carotid Stenosis; Ischemic Attack; Stroke; Bleeding
Keywords: Carotid atherosclerosis; Carotid stenosis; Ischemic attack; Stroke; Carotid stenting; Transradial approach; Transfemoral approach; Bleeding; Thromboembolism; Embolism; Neurocognitive disorders
MeSH Terms: conditions — Carotid Artery Diseases; Carotid Stenosis; Stroke; Hemorrhage; Thromboembolism; Embolism; Neurocognitive Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carotid stenting, Transradial approach (Experimental): Internal carotid artery stenting using transradial arterial approach
  Interventions: Procedure: Transradial carotid artery stenting
- Carotid stenting, Transfemoral approach (Active Comparator): Internal carotid artery stenting using transfemoral arterial approach
  Interventions: Procedure: Transfemoral carotid artery stenting

INTERVENTIONS:
Procedure: Transradial carotid artery stenting — The radial artery is punctured with a trocar. A guidewire is advanced through its lumen, and the trocar is withdrawn. An introducer is passed into the vessel. Then a standard endovascular procedure is carried out under local anesthesia and fluoroscopic control. To prevent cerebral embolism, a protection device is positioned distally of target lesion in internal carotid artery. Then balloon angioplasty of target lesion (if required) is provided. After the angiographic control stent is implanted. After removing all of devices a control angiographic study is provided. Medical therapy includes aspirin(acid acetylsalicylic) 125 - 300 mg/d and plavix (clopidogrel) in dose 300-600 mg prescription before the procedure and heparin sodium injection during the procedure(5000 U iv). After the procedure aspirin(acid acetylsalicylic) in dose 100 mg/d within long period should be prescribed in all the patients, and Plavix (clopidogrel) in dose 75/d should be prescribed within 2 months.
  Arms: Carotid stenting, Transradial approach
Procedure: Transfemoral carotid artery stenting — The common femoral artery is punctured with a trocar. A guidewire is advanced through its lumen, and the trocar is withdrawn. An introducer is passed into the vessel. Then a standard endovascular procedure is carried out under local anesthesia and fluoroscopic control. To prevent cerebral embolism, a protection device is positioned distally of target lesion in internal carotid artery. Then balloon angioplasty of target lesion (if required) is provided. After the angiographic control stent is implanted. After removing all of devices a control angiographic study is provided. Medical therapy includes aspirin(acid acetylsalicylic) 125 - 300 mg/d and plavix (clopidogrel) in dose 300-600 mg prescription before the procedure and heparin sodium injection during the procedure(5000 U iv). After the procedure aspirin(acid acetylsalicylic) in dose 100 mg/d within long period should be prescribed in all the patients, and Plavix (clopidogrel) in dose 75/d should be prescribed within 2 months.
  Arms: Carotid stenting, Transfemoral approach

SUMMARY:
The aim is to compare the safety of using transfemoral and transradial approach in patient undergoing carotid arteries stenting.

DETAILED DESCRIPTION:
The use of transradial approach in carotid arteries stenting can significantly decrease the amount of adverse events associated with transfemoral approach such as bleeding or hematoma. Otherwise providing transradial approach is fraught with technical difficulties of common carotid artery canulation that can result in embolic complications. Taking into account the absence of studies in this area of medicine, providing investigation evaluating parameters of safety for both methodics is very actual.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic patients with internal carotid artery stenosis(>50%)
* Asymptomatic patients with internal carotid artery stenosis(>60%)
* Anatomy of internal carotid artery applicable for stent implantation and use of embolic protection device

Exclusion Criteria:

* Stroke, myocardial infarction or underwent operative treatment within 1 month
* Prior carotid artery stenting
* Cerebral vessels aneurisms/ malformations
* Subclavian artery/ brachiocephalic trunk stenosis
* Contraindications for antiplatelet or/and anticoagulation therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2015-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Cerebral embolism | during 24 hours after carotid artery stenting
  Amount of intraoperative micro- and macroembolic complications evaluated as an occurence of new ipsilateral ischemic lesions estimated due to brain MRI data.

SECONDARY OUTCOMES:
Cerebral embolism | intraoperative
  Amount of intraoperative microembolic signals revealed by transcranial ultrasound Doppler examination.
MACCE | during 30 days after carotid artery stenting
  Major adverse cardiac and cerebrovascular events (MACCE) including: including: All-cause mortality, Myocardial infarction, Stent thrombosis, Clinically indicated Target lesion revascularization, Any target lesion revascularization, Any target vessel revascularization.
Neurocognitive disorders | before and 30 days after carotid artery stenting
  Mini-Mental State Examination (MMSE)
Neurocognitive disorders | before and 30 days after carotid artery stenting
  Rey Auditory Verbal Learning Test (RALVT)
Neurocognitive disorders | before and 30 days after carotid artery stenting
  Grooved Pegboard test
Neurocognitive disorders | before and 30 days after carotid artery stenting
  Boston Naming Test
Neurocognitive disorders | before and 30 days after carotid artery stenting
  Geriatric Depression Scale
Neurocognitive disorders | before and 30 days after carotid artery stenting
  Weschler Test of Adult Reading (WTAR)
Device success | intraoperative
  Device success is defined as achievement of a final residual diameter stenosis 20% during the initial procedure.
Lesion success | intraoperative
  Lesion success, defined as achievement of a final residual diameter stenosis 20% with use of any percutaneous coronary intervention (PCI) approach.
In-hospital procedure success | Within 5-day hospitalization
  Procedure success is defined as achievement of a final residual diameter stenosis 20% together with the absence of any in-hospital major adverse cardiac event.
Operative access complications | intraoperative/ 1 day after operation
  Bleeding, aneurisms, large hematomas, atrioventricular fistula
Fluoroscopic time | intraoperative

CONTACTS AND LOCATIONS:
Locations (1):
- State Research Institute of CIrculation Pathology, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No